CLINICAL TRIAL: NCT03050424
Title: Iron and Chronic Obstructive Pulmonary Disease (COPD) Exercise Trial
Acronym: ICE-T
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016LF003B; 2016-000829-39 (EudraCT Number); 16/EE/0355 (Other: REC Reference)
Record Dates: First submitted 2017-02-07; First posted 2017-02-10 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Iron; Exercise Capacity; Non-anaemic iron deficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo-controlled, randomised trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Ferric Carboxymaltose (FCM) (Ferinject) at 15 mg iron/kg body weight
  Interventions: Drug: Ferric Carboxymaltose
- Placebo (Placebo Comparator): Sodium Chloride 0.9%
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Ferric Carboxymaltose — Ferric Carboxymaltose injectable Product
  Other Names: Ferinject®
  Arms: Active
Drug: Sodium Chloride 0.9% — Sodium Chloride 0.9%
  Arms: Placebo

SUMMARY:
This phase II single centre, double blind, placebo-controlled, randomised trial aims to test the hypothesis that intravenous iron improves exercise performance in Chronic Obstructive Pulmonary Disease (COPD) as measured by constant rate cycle ergometry.

DETAILED DESCRIPTION:
Iron deficiency (ID) is one of the most common nutritional deficiencies affecting humans. Chronic diseases, including COPD, are commonly complicated by iron deficiency anaemia (IDA). It has been well documented that there is an association between both ID and anaemia and reduced exercise capacity. It has been postulated that addressing this ID may be a novel approach to improve exercise capacity and quality of life.

The ECLIPSE cohort found that the prevalence of anaemia in patients with COPD is 19% and is associated with functional limitation and poor outcomes; similarly Nickol et al (2015) found ID to be prevalent in 17.7% of patients with COPD.

Barberan-Garcia et al (2015) evaluated the relationship between Non-anaemic iron deficiency (NAID) and aerobic capacity in seventy COPD patients before and after an 8 week high intensity endurance exercise training programme. Endurance time was assessed as endurance time during constant work rate exercise testing at 80% of oxygen consumption (VO2) peak. At baseline it was noted that the NAID group in comparison to the normal iron status group had a lower exercise tolerance of approximately 90 seconds, which is close to normally reported minimal clinical important difference (MCID's) for this test, P=0.007. After adjusting for confounding variables with a multiple regression analysis it was shown that training induced increase in aerobic exercise capacity was only found in the normal iron status group, with the effect of training on exercise tolerance being lower in the NAID (P=0.041).

Exercise capacity in COPD is strongly linked to outcome measures and mortality. The benefit of correcting NAID in COPD subjects would be to achieve an increase in exercise endurance and thus an improvement in Quality of Life (QoL). Currently there is no standard treatment for NAID in COPD, so this pilot, randomised, double-blind, placebo-controlled trial will attempt to answer this question.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically stable patients (>18 years old), Global Initiative for Chronic Obstructive Lung Disease (GOLD) II-IV COPD Forced Expiratory Volume in 1 second (FEV1):Forced Vital capacity (FVC) < 0.70
2. Non-anaemic: males haemoglobin (Hb) ≥ 130g/L, and females ≥ 120g/L
3. Iron deficiency, defined as:

   1. Serum Ferritin < 100 µg/ml
   2. Serum Ferritin 100-299 µg/ml with Transferrin saturation (TSAT) < 16%
   3. Soluble transferring receptor > 28.1nmol/L
4. No history of lower respiratory tract infection or exacerbation of COPD in the last 6 weeks
5. No participation in Pulmonary Rehabilitation (PR) for at least 3 months prior to initial assessment.

Exclusion Criteria:

1. Polycythemia defined as Hb > 170g/L and haematocrit > 0.6 in males and Hb > 150g/L and haematocrit > 0.56 in females.
2. Significant co-morbidity contributing to reduced exercise tolerance
3. Congestive cardiac failure defined as Left Ventricular Ejection Fraction (LVEF) < 45% or plasma B-type natriuretic peptide (BNP) > 100pg/ml.
4. Oral iron therapy at doses > 100mg/day in the previous week prior to randomisation.
5. Chronic liver disease (including active hepatitis) and/or screening alanine transaminase or aspartate transaminase above 3 times the upper limit of normal range.
6. Anaemia (WHO [31]) defined as Hb < 130g/L in males > 15 yrs old and Hb < 120g/L in non-pregnant females.
7. Current malignancy or haematological disorders.
8. Currently receiving systemic chemotherapy and/or radiotherapy.
9. Renal dialysis (previous, current or planned).
10. Unstable angina.
11. Subject is of child-bearing potential or is pregnant or breast feeding.
12. Contraindication to Ferrous Carboxymaltose (Ferinject):

    1. Hypersensitivity to active substance
    2. Known serious hypersensitivity to other parental iron substance
    3. Anaemia not attributed to iron deficiency (e.g. other microcytic anaemia)
    4. Evidence of iron overload or disturbance in utilisation of iron.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Constant Rate Cycle Ergometry (75% Max Load) | 8 weeks
  Increased exercise capacity as assessed by endurance cycle ergometry at 75% VO2max

SECONDARY OUTCOMES:
Quality of Life | Week 0; Week 8; Week 10; Week 14
  COPD Assessment Test (CAT)
Quality of Life | Week 0; Week 8; Week 10; Week 14
  Medical Research Council (MRC) Dyspnoea Scale
Quality of Life | Week 0; Week 8; Week 10; Week 14
  Hospital Anxiety and Depression (HAD) Scale
Quality of Life | Week 0; Week 8; Week 10; Week 14
  Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F)
Quality of Life | Week 0; Week 8; Week 10; Week 14
  EuroQoL Group (EQ-5D-5L)
Muscle Oxygen Delivery | Week 0; Week 8; Week 14
  Near infrared spectroscopy during muscle contraction
Endurance Shuttle Walk Test (ESWT) | Week 0; Week 4; Week 10; Week 14
  Change in endurance shuttle walk test distance and time
Adverse Effects of Iron Administration | Week 0; Week 4; Week 8; Week 10; Week 14
  Any adverse effects of intravenous iron administration

CONTACTS AND LOCATIONS:
Overall Officials: Michael Polkey, MRCP, PhD, Principal Investigator — Royal Bromtpon and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demeyer H, Louvaris Z, Frei A, Rabinovich RA, de Jong C, Gimeno-Santos E, Loeckx M, Buttery SC, Rubio N, Van der Molen T, Hopkinson NS, Vogiatzis I, Puhan MA, Garcia-Aymerich J, Polkey MI, Troosters T; Mr Papp PROactive study group and the PROactive consortium. Physical activity is increased by a 12-week semiautomated telecoaching programme in patients with COPD: a multicentre randomised controlled trial. Thorax. 2017 May;72(5):415-423. doi: 10.1136/thoraxjnl-2016-209026. Epub 2017 Jan 30. PMID 28137918
- [Background] Zoumot Z, Davey C, Jordan S, McNulty WH, Carr DH, Hind MD, Polkey MI, Shah PL, Hopkinson NS. Endobronchial valves for patients with heterogeneous emphysema and without interlobar collateral ventilation: open label treatment following the BeLieVeR-HIFi study. Thorax. 2017 Mar;72(3):277-279. doi: 10.1136/thoraxjnl-2016-208865. Epub 2016 Dec 20. PMID 27999170
- [Background] Nolan CM, Maddocks M, Canavan JL, Jones SE, Delogu V, Kaliaraju D, Banya W, Kon SSC, Polkey MI, Man WD. Pedometer Step Count Targets during Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2017 May 15;195(10):1344-1352. doi: 10.1164/rccm.201607-1372OC. PMID 27911566
- [Background] Demeyer H, Gimeno-Santos E, Rabinovich RA, Hornikx M, Louvaris Z, de Boer WI, Karlsson N, de Jong C, Van der Molen T, Vogiatzis I, Janssens W, Garcia-Aymerich J, Troosters T, Polkey MI; PROactive consortium. Physical Activity Characteristics across GOLD Quadrants Depend on the Questionnaire Used. PLoS One. 2016 Mar 14;11(3):e0151255. doi: 10.1371/journal.pone.0151255. eCollection 2016. PMID 26974332
- See also: Drug information for Sodium Chloride Injection BP 0.9% w/v — https://www.medicines.org.uk/emc/medicine/20890
- See also: Drug information for Ferinject (ferric carboxymaltose) — https://www.medicines.org.uk/emc/medicine/24167